CLINICAL TRIAL: NCT04675853
Title: Rapid dEvice Testing pROtocol for Parkinson's Disease (RETRO-PD)
Brief Title: Rapid dEvice Testing pROtocol for Parkinson's Disease
Acronym: RETRO-PD
Status: Completed | Type: Observational
Sponsor: HealthMode Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HM041001
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Healthy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PD
- Care Partners of PD participants

SUMMARY:
This is an 8 week observational study to evaluate the feasibility of using remote monitoring technologies in future studies of PD. The study will 2 clinical evaluations (one initial, one final), and an 8-week monitoring period including 4 virtual visits where participants will use a combination of digital devices (Emerald touchless sensor system with associated ankle accelerometer, iPhone, Apple Watch, iPad, Fitbit Aria, FitBit Versa, Withings Blood Pressure Monitor Connect, and/or Withings Sleep Mat) during their daily lives.

ELIGIBILITY:
Inclusion Criteria:

Participants with PD

* At least 30 years of age
* Clinical diagnosis of PD by a neurologist or other movement disorder specialist as reported by the participant, with current motor symptoms
* Able to ambulate independently (assistance of minor walking aids such as a cane is permitted, but depending on a walker for ambulation is not)
* Have a BMI of 33 or below calculated by participant reported height and weight at the time of screening
* Have a care partner who meets the study's inclusion criteria
* Able to read, understand, and provide written informed consent in English
* Able, either alone or with a care partner, to operate digital devices
* Have reliable wifi in their home and the ability to connect new devices to their home wifi

Care partners

* At least 18 years of age
* Able to read, understand, and provide written informed consent in English
* Able to operate digital devices
* Care partner for the participant with PD enrolled in the study
* Lives with the participant with PD enrolled in the study
* Able to ambulate independently (assistance of minor walking aids such as a cane is permitted, but depending on a walker for ambulation is not)
* Willing to exclude pet from the participant's bedroom at night for the duration of the study

Exclusion Criteria:

Participants with PD

* Any non-PD forms of Parkinsonism
* Active psychiatric disorders that affect the ability to complete study tasks
* Any other medical condition that is the primary cause of the present movement disorder
* Cognitive dysfunction (score > 7 on the Six-Item Cognitive Impairment Test)
* Considered by the investigator to be an unsuitable participant
* Live in a household with more than three people
* Unwilling to exclude pet from their bedroom at night for the duration of the study

Care partners

* Cognitive dysfunction (score > 7 on the Six-Item Cognitive Impairment Test)
* Considered by the investigator to be an unsuitable participant

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll at least 25 dyads consisting of participants with PD and their care partners recruited from multiple clinical practices and the general public. Participants who withdraw from the study before completing virtual visit V04 (day 28) will be replaced. Enrollment will be enriched to ensure that participants are distributed across mild to severe PD.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
The feasibility of digital and remote monitoring technologies | 8 weeks
  determined by evaluating:
  1. Ease of deployment and initial set-up, utility of technology and user experience as reported by the usability surveys and interview questionnaires (measured by means of Standard Usability Questionnaire score ranges from 10 to 50, higher score indicating a better usability)
  2. Total time and percentage of continuous data collection for each stream of data and frequency and distribution of missing data points.
  3. Mutual consistency of data from multiple, related data streams
  4. Data utility reports
  5. Responses from participants with PD and care partners regarding ease of use and comfort of technologies in study
  6. Adherence of participants to active tasks and use of the devices

SECONDARY OUTCOMES:
Correlation with standard measures | 8 weeks
  Correlation of data from the included digital technologies and their relationship to standard measures (correlations with scores from MDS-UPDRS, PDQ-8 and SE-ADL)

CONTACTS AND LOCATIONS:
Locations (1):
- Mobile Clinical Research Site, New York, New York, United States